CLINICAL TRIAL: NCT07338487
Title: A Prospective, Randomized, Parallel-Controlled Clinical Study of Nanocrystalline Megestrol Acetate in Concurrent Chemoradiotherapy for Locally Advanced Cervical Cancer
Brief Title: A Clinical Study of Nanocrystalline Megestrol Acetate in Concurrent Chemoradiotherapy for Locally Advanced Cervical Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Jingjing Wang, associate chief physician, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LYEC2024-0342
Record Dates: First submitted 2025-12-14; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Cervical Cancer; Cachexia
Keywords: Locally Advanced Cervical Cancer; Nanocrystalline Megestrol Acetate; Cachexia; Clinical Research; Control Group
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nanocrystalline Megestrol Acetate Oral Suspension (Experimental)
  Interventions: Drug: Nanocrystalline Megestrol Acetate Oral Suspension
- Placebo Control (No Intervention)

INTERVENTIONS:
Drug: Nanocrystalline Megestrol Acetate Oral Suspension — Nanocrystalline Megestrol Acetate Oral Suspension, 125 mg/mL specification, administered orally at 5 mL (625 mg/day) daily in the study arm for a duration of 8 weeks.
  Arms: Nanocrystalline Megestrol Acetate Oral Suspension

SUMMARY:
Cervical cancer, ranking as the fourth most prevalent malignancy in women globally, presents significant challenges in nutritional management. Approximately 31% of patients develop cancer-related malnutrition/cachexia, with 10-20% of deaths directly attributable to nutritional depletion. The disease process and its treatment - particularly concurrent chemoradiotherapy (CCRT) - create a destructive cycle through multiple mechanisms. Tumor-derived factors (including activins and myostatin) and inflammatory cytokines (such as TNF-α and IL-6) actively promote muscle and fat catabolism. CCRT toxicity, especially from platinum-based drugs, worsens this condition by inducing mitochondrial dysfunction and accelerating protein degradation, leading to clinically significant sarcopenia. This metabolic disruption has dire consequences, with studies showing severe weight loss during CCRT correlating with a 2.37-fold increase in mortality risk (HR 2.37, p=0.036).

Nanocrystalline megestrol acetate (MA) emerges as a promising therapeutic intervention with dual mechanisms of action. Centrally, it modulates D2 receptors to upregulate neuropeptide Y (NPY), effectively stimulating appetite. Peripherally, it suppresses key inflammatory cytokines (IL-6 and TNF-α), thereby reducing systemic inflammation and muscle wasting. Its efficacy is well-established, with endorsement from major oncology guidelines (ASCO, NCCN, ESMO) for cancer cachexia management. A comprehensive meta-analysis of 35 clinical trials involving 4,234 patients demonstrated MA's superiority over placebo, showing significant improvements in appetite (RR 2.2), weight gain (RR 1.6), and quality of life (RR 1.8).

The nanocrystalline formulation represents a substantial pharmacological advancement over conventional MA. While traditional preparations have limited solubility (2 µg/mL) and require high-fat meals for adequate absorption, the nanocrystalline version (with particles reduced to 26.6 nm) demonstrates 22% greater bioavailability. This translates to clinically meaningful differences: fasting-state peak concentrations increase from 187 ng/mL to 1,133 ng/mL, the time to observable effect shortens from 14 days to just 3 days, and 12-week weight gain improves from 3.5 kg to 5.4 kg (with 40% being lean mass). Dose optimization studies confirm 800 mg/day as the optimal conventional MA dose, with the nanocrystalline equivalent being 625 mg/day due to its enhanced bioavailability.

The proposed clinical investigation will evaluate this intervention in FIGO IB3-IVA cervical cancer patients (n=5) undergoing CCRT. The study employs a two-arm design comparing nanocrystalline MA (625 mg/day) plus CCRT against CCRT alone. Primary endpoints focus on BMI changes at 8 weeks, with secondary assessments of nutritional status, inflammatory markers, and quality of life measures. This research aims to establish nanocrystalline MA as a means to break the cachexia cycle in cervical cancer treatment, potentially improving both treatment tolerance and survival outcomes.

ELIGIBILITY:
Eligibility Criteria:

1. Voluntarily sign the written ICF.
2. Age ≥ 18 years at the time of enrollment.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
4. Expected survival period ≥ 6 months.
5. Histologically or cytologically confirmed locally advanced cervical cancer (Stage IB3/IIA2/IIB-IVA) that is not amenable to complete surgical resection, classified according to the International Federation of Gynecology and Obstetrics (FIGO) staging system.
6. Scheduled to undergo radical concurrent chemoradiotherapy.
7. At least one measurable tumor lesion according to RECIST v1.1.
8. Adequate organ function defined as follows:

   a) Hematology (without any blood component or growth factor support within 7 days prior to initiation of study treatment): i. Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L (1,500/mm³); ii. Platelet count ≥ 100 × 10⁹/L (100,000/mm³); iii. Hemoglobin ≥ 90 g/L. b) Renal: i. Calculated creatinine clearance* (CrCl) ≥ 50 mL/min
   * CrCl will be calculated using the Cockcroft-Gault formula:

   CrCl (mL/min) = (140 - age) × weight (kg) × F / (serum creatinine [mg/dL] × 72) F = 1 for males; F = 0.85 for females ii. Urine protein ≤ 1+ or 24-hour urinary protein quantification < 1.0 g. c) Hepatic: i. Total bilirubin (TBil) ≤ 1.5 × ULN; for patients with liver metastases or confirmed/suspected Gilbert's disease, TBil ≤ 3 × ULN; ii. AST and ALT ≤ 2.5 × ULN; for patients with liver metastases, AST and ALT ≤ 5 × ULN; iii. Serum albumin (ALB) ≥ 28 g/L. d) Coagulation: i. International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (unless the patient is receiving anticoagulant therapy and coagulation parameters [PT/INR and APTT] are within the therapeutic range at screening).

   e) Cardiac: i. Left ventricular ejection fraction (LVEF) ≥ 50%.
9. Female patients of childbearing potential must have a negative urine or serum pregnancy test within 3 days prior to the first dose (if urine pregnancy test result is not confirmed negative, a serum pregnancy test will be required, and the serum result shall prevail). If a female patient of childbearing potential engages in sexual activity with a non-sterilized male partner, she must use acceptable contraceptive methods starting from screening and continue for 120 days after the last dose of study drug; whether to discontinue contraception after this time point should be discussed with the investigator. If a non-sterilized male patient engages in sexual activity with a female partner of childbearing potential, he must use effective contraceptive methods from screening until 120 days after the last dose; whether to discontinue contraception after this time point should be discussed with the investigator.
10. The patient is willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study requirements.

Exclusion Criteria:

Patients meeting any of the following criteria will be ineligible for this study:

1. Conditions affecting gastrointestinal absorption such as dysphagia, malabsorption, or uncontrolled vomiting; ongoing tube feeding or parenteral nutrition; presence of anorexia nervosa, psychogenic anorexia, or pain-induced feeding difficulties.
2. Current or planned use of medications that increase appetite or weight, including but not limited to: adrenal corticosteroids (except short-term dexamethasone during chemotherapy), androgens, progestins, thalidomide, olanzapine, anamorelin, or other appetite stimulants.
3. Diagnosis of Cushing's syndrome, adrenal or pituitary insufficiency; poorly controlled diabetes mellitus.
4. Current radiographic or clinical evidence of gastrointestinal obstruction.
5. Active autoimmune disease requiring systemic treatment within the past two years (e.g., disease-modifying agents, corticosteroids, immunosuppressants). History of non-infectious pneumonitis/interstitial lung disease requiring systemic glucocorticoid therapy, or current non-infectious pneumonitis.
6. Uncontrolled concurrent illnesses including but not limited to decompensated cirrhosis, renal failure, uncontrolled metabolic disorders, severe active peptic ulcer disease/gastritis, or psychiatric/social conditions that would limit compliance with study requirements or the ability to provide written informed consent.
7. Within 12 months prior to the first dose: unstable angina requiring hospitalization, myocardial infarction, congestive heart failure (NYHA Class II or higher), vascular disease (e.g., aortic aneurysm at risk of rupture), or other cardiac impairments that may affect safety evaluation of the study drug (e.g., poorly controlled arrhythmia, myocardial ischemia). Within 6 months prior to the first dose: history of esophagogastric varices, severe ulcers, gastrointestinal perforation and/or fistula, gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), intra-abdominal abscess, or acute gastrointestinal bleeding.
8. Within 6 months prior to the first dose: any arterial thromboembolic events, Grade 3 or higher venous thromboembolism per NCI CTCAE v5.0 requiring urgent intervention (e.g., pulmonary embolism or intracardiac thrombosis), transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy. Within 1 month prior to the first dose: acute exacerbation of chronic obstructive pulmonary disease. Current hypertension with systolic BP ≥160 mmHg or diastolic BP ≥100 mmHg despite oral antihypertensive therapy.
9. History of severe bleeding tendency or coagulopathy; clinically significant bleeding symptoms within 1 month prior to the first dose, including but not limited to gastrointestinal bleeding, hemoptysis (defined as coughing/expectorating ≥1 teaspoon of fresh blood or small clots, or blood without sputum; patients with blood-tinged sputum are eligible), epistaxis (excluding minor nasal bleeding and blood-tinged postnasal drip).
10. Within 4 weeks prior to the first dose: severe infections including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia; within 2 weeks prior to the first dose: active infection requiring systemic antimicrobial therapy (excluding antiviral therapy for hepatitis B/C).
11. Any condition, treatment, or laboratory abnormality that may confound study results, impede complete study participation, or make participation not in the patient's best interest.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate the change in BMI during concurrent chemoradiotherapy with Nanocrystalline Megestrol Acetate in locally advanced cervical cancer. | Treatment shall continue until disease progression or for up to 8 weeks (maximum treatment duration: 8 weeks).

SECONDARY OUTCOMES:
Change in appetite score as measured by the AC/S-12 scale over an 8-week period. | Treatment shall continue until disease progression or for up to 8 weeks (maximum treatment duration: 8 weeks)
To evaluate the progression-free survival (PFS) rate of Nanocrystalline Megestrol Acetate during concurrent chemoradiotherapy for locally advanced cervical cancer (assessed per RECIST v1.1). | Treatment shall continue until disease progression or for up to 8 weeks (maximum treatment duration: 8 weeks)
To assess lean body mass change with Nanocrystalline Megestrol Acetate | Treatment shall continue until disease progression or for up to 8 weeks (maximum treatment duration: 8 weeks)
To assess treatment cycle completion rates with Nanocrystalline Megestrol Acetate | Treatment shall continue until disease progression or for up to 8 weeks (maximum treatment duration: 8 weeks)
To evaluate the incidence and severity of radiotherapy-related adverse events | Treatment shall continue until disease progression or for up to 8 weeks (maximum treatment duration: 8 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Second Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided